CLINICAL TRIAL: NCT05837767
Title: A Pilot Study of Spatially Fractionated Radiation Therapy in Patients With Extra-Cranial Soft Tissue Metastases
Brief Title: A Study of Radiation Therapy to Treat Solid Tumor Cancer That Has Spread to Soft Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-207
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Invasive Ductal Breast Carcinoma; Invasive Ductal Breast Carcinoma Stage IV; Lobular Breast Carcinoma; Lobular Breast Carcinoma Stage IV; Non Small Cell Lung Cancer; NSCLC; Gastrointestinal Cancer; Gastrointestinal Squamous Cell Cancer; Gastrointestinal Adenocarcinoma; Pancreatic Cancer; Bladder Cancer; Renal Cell Carcinoma; Melanoma; Sarcoma; Metastatic Solid Tumor
Keywords: Invasive Ductal Breast Carcinoma; Lobular Breast Carcinoma; Non Small Cell Lung Cancer; NSCLC; Gastrointestinal Cancer; Gastrointestinal Squamous Cell Cancer; Pancreatic Cancer; Bladder Cancer; Renal Cell Carcinoma; Melanoma; Sarcoma; Metastatic Solid Tumor; extra-cranial disease; lattice radiation therapy; LRT; spatially fractionated radiation therapy; SFRT; SBRT; stereotactic body radiation therapy; 22-207; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Carcinoma, Lobular; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Melanoma; Sarcoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with metastatic solid tumors (Experimental): Participants will have metastatic solid tumors and at least two sites of measurable extra-cranial disease
  Interventions: Radiation: Palliative radiotherapy

INTERVENTIONS:
Radiation: Palliative radiotherapy — Palliative radiotherapy (RT) will be performed using external beam ionizing radiation in accordance with standard practice

SUMMARY:
The purpose of this study is to find out whether lattice radiation therapy (LRT) is an effective radiation therapy technique when compared to standard stereotactic body radiation therapy (SBRT). The study will also study how the different radiation therapy techniques (LRT and SBRT) affect how many immune cells are able to attack and kill tumor cells (immune infiltration).

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy confirmed advanced/metastatic solid tumors of the following types: invasive ductal or lobular breast carcinoma (all histological and intrinsic subtypes), non-small cell lung cancer (NSCLC, all subtypes), gastrointestinal squamous cell or adenocarcinomas (including pancreatic cancer), bladder cancer, renal cell carcinoma, melanoma, and soft tissue sarcoma (all subtypes), who require and are being planned for palliative radiation therapy to at least one site of extracranial metastatic disease measuring at least 5 cm in a single axis. If a patient, requires palliative radiotherapy to additional sites, these can be treated with standard of care SBRT per departmental guidelines.
* Age ≥ 18 years
* ECOG Performance Status of 0 or 1.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Prior radiation therapy to the candidate metastatic sites under consideration for treatment ("re-irradiation" is disallowed).
* Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus, or connective tissue diseases (lupus, systemic sclerosis, or other collagen vascular diseases) that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Patients with a "currently active" metastatic second malignancy.
* Patients on oral or parental corticosteroids. Physiological doses of steroids are permitted (eg for patients with adrenal insufficiency). If patients are on supraphysiological doses of steroids, these must be discontinued and held during the period of the study.
* Concomitant anti-neoplastic treatment is not allowed during the days of radiation treatment delivery and should be completed or held for 3 days prior to commencement of protocol treatment and for 3 days following completion of radiotherapy, or with resolution of associated acute toxicities.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 12 weeks from baseline
  The primary endpoint is ORR in the LRT-treated lesion, as defined by RECIST v.1.1 criteria, at 12 weeks on a standard-of-care response assessment CT or F-18-FDG PET/CT scan after LRT.

CONTACTS AND LOCATIONS:
Overall Officials: Atif Khan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org